CLINICAL TRIAL: NCT04472845
Title: HYPofractionated Adjuvant RadioTherapy in 1 Versus 2 Weeks in High-risk Patients With Breast Cancer (HYPART): A Non-inferiority, Open-label, Phase III Randomized Trial.
Brief Title: HYPofractionated Adjuvant RadioTherapy in 1 Versus 2 Weeks in High-risk Patients With Breast Cancer (HYPART).
Acronym: HYPART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPART
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Hypofractionation; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 week (Experimental): Radiotherapy dose to chest wall, axilla level III and supraclavicular fossa will be of 26Gy in 5 fractions over 1 week in the study arm. BCS patients will receive a sequential boost of 8Gy/2#/2days or simultaneous integrated boost(SIB) to a total dose of 34Gy.Supraclavicular fossa(SCF) and axilla level III will be treated in patients with T3-4 disease with lymphovascular invasion, grade 3 or N2 disease and T3-4 disease treated with neoadjuvant chemotherapy after adequate axillary dissection. Level I and II axilla will only be irradiated in patients with inadequate axillary dissection(<10 lymph nodes). Internal mammary node (IMNs) radiation will be done in T3-4 central and inner quadrant lesions and patients with N2 disease. IMNs will be irradiated with a separate single field. The first five intercostal spaces will be included in the IMN target volume.
  Interventions: Radiation: 1 week RT
- 2 week (Active Comparator): Radiotherapy dose to chest wall, axilla level III and supraclavicular fossa will be 34Gy in 10 fractions over 2 weeks in the control arm. BCS patients will receive a sequential boost of 8Gy/2#/2days or simultaneous integrated boost(SIB) to a total dose of 42 Gy.
  Interventions: Radiation: 2 week RT

INTERVENTIONS:
Radiation: 1 week RT — RT will be delivered over 1 week
  Arms: 1 week
Radiation: 2 week RT — RT will be delivered over 2 week
  Arms: 2 week

SUMMARY:
We at PGIMER have been practicing hypofractionated radiotherapy in breast cancer patients for the last 4 decades. Our standard doses have been 35Gy/15#/3wks to the chest wall after mastectomy and 40Gy/16#/3wks after breast conserving surgery (BCS).It is also a routine practice in the UK and in a few centers in Canada. Hypofractionation reduces treatment time to half while maintaining cosmesis and gives control rates equal to conventional fractionation. As breast cancer is a leading cancer in females and radiation therapy is an important part of its local management, hypofractionation helps radiation centers worldwide to meet the growing need for radiation treatment in breast cancer, particularly in developing countries where resources are limited. It also reduces the financial burden on the patient and family. In this study we want to evaluate the impact of reducing the treatment duration from 3 weeks to 1 week. Eligible patients with breast cancer after mastectomy or BCS will be treated with a radiotherapy dose of 26Gy in 5 fractions over 1 week in the study arm and 40Gy in 15 fractions over 2 weeks in the control arm. The primary endpoint of this noninferiority study will be locoregional tumour control. Secondary endpoints will be early and late radiation toxicities, quality of life, contralateral primary tumours, regional and distant metastases, survival and second cancers. A total of 1018 patients will be randomised (1:1) to receive 1 week or 2 weeks of radiotherapy. An event-driven analysis will be performed after at least 94 patients have documented locoregional recurrences.

DETAILED DESCRIPTION:
Aim: To test a 1-week schedule of hypofractionated adjuvant whole breast/chest wall and/or regional nodal radiotherapy against 2 weeks for loco-regional control, acute and late toxicities, quality of life (QoL), survival and second cancers after primary surgery in patients with breast cancer.

Review of literature Four randomised trials involving a total of >8000 women have compared a lower total dose in fewer larger fractions against 50Gy in 25 fractions, and all have reported favourable results in terms of local tumour control and late adverse effects.1-4 Appropriate adjustments to total dose allow 15- or 16-fraction schedules to be delivered over 3 weeks that are at least as safe and effective as standard 5-week regimens.

A 2008 Cochrane review of altered radiotherapy fractionation in early breast cancer1 including The Royal Marsden Hospital/Gloucestershire Oncology Centre and Ontario trials totalling 2644 women with mainly axillary node negative tumours <5cm diameter concluded that radiotherapy fractions larger than 2Gy were at least as effective as 2Gy fractionation for a) local-recurrence free survival (absolute difference 0.4%, 95% CI 1.5% to 2.4%), b) breast appearance (risk ratio (RR)1.01, 95% CI 0.88 to 1.17; p=0.86), c) survival at five years (RR 0.97, 95% CI 0.78 to 1.19; p=0.75), d) late skin toxicity at five years (RR 0.99, 95% CI 0.44 to 2.22; p=0.98, or e) late radiation toxicity in subcutaneous tissue (RR1.0, 95% CI 0.78 to 1.28; p=0.99).1 The UK START A trial(N=2236) showed that the estimated absolute differences in 5-year local-regional relapse rates compared with the control schedule of 50Gy in 2Gy fractions were 0.2% (95% CI 1.3% to 2.6%) after41.6Gy and 0.9% (95% CI 0.8% to 3.7%) after 39Gy. In STARTA, photographic and patient self- assessments suggested lower rates of late adverse effects after 39 Gy than with 50 Gy, with a hazard ratio(HR) for late change in photographic breast appearance of 0.69(95% CI 0.52 to 0.91,p=0.01).3 In the UK START B trial(N=2215) the estimated absolute difference in 5-year local-regional relapse rates for 40.05 Gy compared with 50Gy was -0.7% (95% CI 1.7% to 0.9%),and the HR for late change in photographic breast appearance was 0.83 (95% CI 0.66 to1.04). These START trials reported similar local tumour control with some evidence of lower rates of late adverse effects after schedules with fraction sizes larger than 2 Gy compared with the international standard 25-fraction regimen.4 The international standard regimen for whole breast radiotherapy prior to publication of these studies was a total dose of 50Gy in 25 fractions (daily doses) over 5weeks following surgical resection of the primary tumour in women with early breast cancer. With the establishment of safety and efficacy of moderate hypofractionation another 'new standard of care' using 40-41Gy in 15 to 16 fractions over 3 weeks has been established, as evidenced by recommendations by the National Institute for Health and Clinical Excellence(NICE). 5 Although interesting and practically helpful, such moderate hypofractionation is unlikely to represent the useful limits of hypofractionation for whole breast or even regional nodal radiotherapy.

Further hypofractionated radiotherapy has been tested using once weekly schedule to the whole breast in the UK FAST study.5 Assuming an α/β value between 3 and 4 two different schedules were hypothesised to be equally effective (28.5 Gy and 30Gy in 5 fractions over 5 weeks) to the 50Gy in 25 fraction over 5 weeks schedule. Initial analysis has shown a higher rate of moist desquamation using the 50Gy regimen; however photographic assessment after a median follow-up of 28.4 months has shown more mild or marked change in the photographic appearance with the hypofractionated schedule.4 Clinical assessments of breast appearance changes were similar to the 50Gy group when using the 28.5Gy schedule but worse with the 30Gy schedule. Final results from the study are awaited. The UK FAST Forward study randomly allocated 4096 patients to 40Gy/15#/3 weeks, 27Gy/5#/1 week, or 26Gy/5#/1 week to the whole breast or chest wall.6 They concluded that 26Gy/5#/1 week was non-inferior to the standard of 40Gy/15#/3 weeks for local tumour control, and was as safe in terms of normal tissue effects up to 5 years in patients with early-stage breast cancer.

Hypofractionated radiotherapy has been used at PGIMER and comparable clinical outcomes have been published with moderate hypofractionation.7-9 Although Indian breast cancer patients present at a younger age, with more advanced stage, and a higher percentage of grade 3 and triple negative tumours compared to the western population. These adverse factors may not be important when comparing hypofractionated radiotherapy with standard fractionation.9 Reservations exist for extreme hypofractionation to the regional nodes citing increasing risk of brachial plexopathy when hypofractionating to the supraclavicular fossa although moderate hypofractionation has been used at our institute for the last 5 decades without reports of any brachial plexopathy.10,11 Similarly, moderately hypofractionated 2-week regimes have been used in clinical trials and have been found to be safe.10 Given the above evidence, 40Gy in 15 fractions has been recommended as the standard of care in the UK even for cases that will include irradiation of the supraclavicular fossa.

Recently, Wang et al. published results from a randomised study in high-risk breast cancer patients after mastectomy.11 They reported similar 5-year clinical outcomes and late toxicities with conventional and hypofractionation. This study also established the safety of 3 weeks regional nodal irradiation(RNI) in patients with breast cancer. They reported a lymphedema rate of 19% at 5-years. We published our results of RNI with 40 Gy/15 fractions/3 weeks hypofractionation with 2D technique, at 15 years RNI was safe and comparable to historical data of conventional fractionation (ClinicalTrial.gov Registration No. NCT04175821).12

Against this background, a phase III randomised, non-inferiority study testing 1 week against 2 weeks of radiotherapy to the breast and chest wall with or without supraclavicular fossa adjuvant radiotherapy will include 1018 patients. The primary end point will be locoregional control and secondary end points will be acute and late radiation toxicity, QoL, survival and second cancers.

5. Preliminary work done: i) The consent form prepared. ii) CRF, PIS, evaluation sheet prepared Detailed Research Methodology This study will be a randomised, non-inferiority, open-label, phase 3 trial, with patients to be recruited from a single institute. Other institutes will be invited if they are willing to participate. Patients to be included in this study will be pre-operatively staged according to American Joint Committee on Cancer (AJCC) 8th edition, International Union against cancer (which uses TNM staging) as stage III breast carcinoma. For patients who receive adjuvant chemotherapy, pathological stage will be reflected and those with neoadjuvant chemotherapy the stage which is higher (clinical/pathological) will be reflected. A total of 1018 patients with histologically proven post lumpectomy/mastectomy cases of carcinoma breast suitable for radiotherapy will be enrolled in this study. Patients will be evaluated at the Department of Radiation Oncology Post Graduate Institute of Medical Education &Research, Chandigarh, India. A thorough clinical examination followed by routine investigations which will include hemogram, liver function tests, kidney function tests, mammography, chest X-ray, ultrasound of abdomen/CECT chest, abdomen and pelvis and whole body bone scan. Written informed consent will be taken from all the patients.

Randomisation and masking Eligible patients will be randomly assigned (1:1) to receive either 1 week or 2 weeks of radiotherapy without stratification by simple randomisation according to a prescribed computer-generated central randomisation schedule. Radiation oncologists in the study team will enroll participants, and research staff members who will be involved in follow-up data collection will assign participants to interventions. Treatment allocation will not be masked.

Radiotherapy Radiotherapy dose to chest wall, axilla level III and supraclavicular fossa will be of 26Gy in 5 fractions over 1 week in the study arm and 34Gy in 10 fractions over 2 weeks in the control arm. BCS patients will receive a sequential boost of 8Gy/2#/2days or simultaneous integrated boost(SIB) to a total dose of 34Gy in the study arm and 42Gy in the control arm. Treatment will be done on a linear accelerator with 6 or 10MV photon energy. Boost can be with photons or electrons. 1cm bolus will be used in all postmastectomy patients, daily in study arm and in 50% of treatment in the control arm. Dose will be prescribed at mid-separation in 2D technique and the dose covering 95% of the planning target volume with three-dimensional conformal(3D-CRT) or intensity modulated radiotherapy(IMRT).

Supraclavicular fossa(SCF) and axilla level III will be treated in patients with T3-4 disease with lymphovascular invasion, grade 3 or N2 disease and T3-4 disease treated with neoadjuvant chemotherapy after adequate axillary dissection. Level I and II axilla will only be irradiated in patients with inadequate axillary dissection(<10 lymph nodes). The prescribed dose to the area will be defined as the dose to the point at 3 cm beneath the skin in two-dimensional radiotherapy technique, or the dose covering 95% of the planning target volume with 3D-CRT or IMRT.

Internal mammary node (IMNs) radiation will be done in T3-4 central and inner quadrant lesions and patients with N2 disease. IMNs will be irradiated with a separate 12x5 cm single field. The first five intercostal spaces will be included in the IMN target volume. The medial border of the IMN field will be midline; lateral border 5 cm lateral to the midline; the superior border will abut the inferior border of the supraclavicular field; and the inferior border will be above the xiphoid. Dose will be 34Gy/10#/2weeks. Dose will be prescribed at 3cm depth. Imaging will be done for set-up verification on alternate days in the study arm and once weekly in the control arm.

Hormonal therapy may be given to oestrogen receptor-positive or progesterone receptor-positive tumours, and anti-HER2-targeted therapy (e.g., trastuzumab) for those with HER2-positive disease depending on the affordability.

Assessment Patients will be assessed for medical history, a physical examination, and a blood test before radiotherapy, once per week during radiotherapy, and 2 weeks after radiotherapy. Patients will be followed up every 3 months for 2 years after radiotherapy, then every 6 months from 3 to 5 years, and yearly thereafter. Skin, subcutaneous toxicity and cosmetic assessment will be done before treatment and then in regular follow up of the study. Acute radiation toxicity will be assessed and scaled according to the RTOG grading system. Late radiation toxicity will be assessed with the Radiation Therapy Oncology Group and the European Organisation for Research and Treatment of Cancer late radiation morbidity scale. Cosmetic assessment will be done using Harvard/NSABP/RTOG breast cosmesis grading scale at baseline, 3 and 5 years. Quality of life(QoL) will be assessed with EORTC QLQ -30, EORTC QLQ-BR 23 at baseline, 3 and 5 years.12

Statistical considerations The primary hypothesis of the study is that locoregional recurrence with 1 week is non-inferior to that with 2 weeks of radiotherapy. The primary endpoint will be locoregional recurrence (LRR). Based on historical data (Wang et al.), the 5-year LRR rate with 3 weeks of RT is expected to be approximately 8%. 1 week RT would be considered non-inferior to 2 weeks RT if the 5-year LRR rate does not exceed 13%. If LRR follows exponential distributions within each treatment group, this non-inferiority margin corresponds to a hazard ratio (HR) of 1.67.

Sample size calculations were performed using module STE0S-3 of nQuery version 8.5.2.0. A total of 94 LRR events will be required to provide at least 80% power using a one-sided test at the 5% level of significance. Under assumed failure rates and guarding against 10% ineligibility or loss to follow-up, the target accrual will be 1018 patients with an accrual period of 3 years. If the two schedules are equivalent, 5 years of follow-up after the last patient has been randomised will be required to observe 94 LRR events, resulting in total study duration of 8 years.

For the primary efficacy endpoint, we will use the cumulative incidence method to estimate the actual incidence of locoregional recurrence at different time points, with death without locoregional recurrence as a competing risk. We will use the log-rank test and Cox regression model for statistical inference based on cause-specific hazards. We will calculate overall survival and disease-free survival using the Kaplan-Meier method, and we will analyse these endpoints using the log rank test and Cox regression model. Acute and late toxicities will be summarised as frequency and severity on the basis of their association with protocol treatment; χ² tests will be used to compare the differences. The primary endpoint and all efficacy endpoints will be analysed in a modified intention-to-treat population (i.e., including all eligible patients who will undergo randomisation but exclude those who are considered ineligible. On the basis of the study design, the primary endpoint locoregional recurrence will be analysed at a one-sided significance level of 0•05 and reported with a two-sided 90% CI. All other statistical tests will be two sided, and p values of <0.05 will be taken as significant. All tests will be performed using SPSS (Statistical Package for the Social Sciences) v.23.0.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Female or male
3. Invasive carcinoma of the breast
4. Breast conserving surgery(BCS) with axillary clearance or total mastectomy with axillary clearance(TMAC); (reconstruction allowed but not with implant; tissue expanders with distant metal ports are allowed)
5. Concurrent trastuzumab and hormone therapy is allowed
6. Axillary staging and/or dissection
7. Complete microscopic excision of primary tumour
8. pT3-4pN2-3 M0 disease
9. Clinical stage III disease or pathological node positive if they have received neo-adjuvant chemotherapy.
10. Written informed consent
11. Able to comply with follow-up

Exclusion Criteria:

1. Supraclavicular node or internal mammary node or distant metastasis
2. Past history of malignancy except (i) basal cell skin cancer and CIN cervix uteri or(ii) non-breast malignancy allowed if treated with curative intent and at least 5 years disease free
3. Contralateral breast cancer, including DCIS, irrespective of date of diagnosis
4. Breast reconstruction using implants
5. Pregnancy
6. Concurrent cytotoxic chemotherapy(sequential neoadjuvant or adjuvant cytotoxic therapy allowed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with conformed invasive breast cancer
Enrollment: 1018 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2028-08-20 (Estimated)

PRIMARY OUTCOMES:
Loco-regional recurrence, Change is being assessed | 5, 10 and 15 years
  disease recurrence in the ipsilateral chest wall or regional lymph nodes from the time of randomization until the end of follow-up.

SECONDARY OUTCOMES:
Disease-free survival, Change is being assessed | 5, 10 and 15 years
  locoregional recurrence, distant metastasis, or death from any cause from the time of randomisation until the end of follow-up.
Overall survival, Change is being assessed | 5, 10 and 15 years
  death from any cause from the time of randomisation until the end of follow-up
Acute radiation toxicity | 3 months
  Any loco-regional toxicity assessed and scaled according to the RTOG grading system.
Late adverse events, Change is being assessed | 5, 10 and 15 years
  Any adverse event occurring after 6 months of RT
Quality of life(QoL), Change is being assessed | Baseline, 3 and 5 years
  QoL will be assessed with EORTC QLQ -30. The QLQ-C30 is composed of both multi-item scales and single-item measures, as well as five functional scales, three symptom scales, a global health status/QoL scale, and six single items. The scores must be averaged and linearly transformed to obtain a range of scores from 0 to 100, with a higher score representing a greater response level.

CONTACTS AND LOCATIONS:
Overall Officials: BUDHI S YADAV, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Budhi Singh Yadav, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadav BS, Sharma SC, Singh R, Singh G, Kumar V. Postmastectomy radiation and survival in patients with breast cancer. J Cancer Res Ther. 2007 Oct-Dec;3(4):218-24. doi: 10.4103/0973-1482.38997. PMID 18270397
- [Background] Yadav BS, Sharma SC, Singh R, Singh G. Patterns of relapse in locally advanced breast cancer treated with neoadjuvant chemotherapy followed by surgery and radiotherapy. J Cancer Res Ther. 2007 Apr-Jun;3(2):75-80. doi: 10.4103/0973-1482.34683. PMID 17998727
- [Background] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Derived] Yadav BS, Goyal S, Dahiya D, Vias P, Gupta A, Datta A, Kataria V, Singh NR, Sharma R, Laroiya I, Irrinki S, P K, Pandey A. HYPofractionated Adjuvant RadioTherapy in 1 Versus 2 Weeks in High-Risk Patients With Breast Cancer (HYPART): Acute Toxicity Results. Int J Radiat Oncol Biol Phys. 2026 Jan 1;124(1):133-146. doi: 10.1016/j.ijrobp.2025.07.1447. Epub 2025 Aug 6. PMID 40780546
- [Derived] Yadav BS, Dahiya D, Kannan P, Goyal S, Laroiya I, Irrinki S, Singh NR, Sharma R. HYPofractionated Adjuvant RadioTherapy in 1 versus 2 weeks in high-risk patients with breast cancer (HYPART): a non-inferiority, open-label, phase III randomised trial. Trials. 2024 Jan 2;25(1):21. doi: 10.1186/s13063-023-07851-7. PMID 38167339